CLINICAL TRIAL: NCT05468294
Title: Phase I/IIb Study of the Tumor Targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With the Anti-PD1 Antibody Nivolumab in Patients With Non-small Cell Lung Cancer
Brief Title: F16IL2 in Combination With Nivolumab in Patients With Non-small Cell Lung Cancer
Acronym: Nivokin
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16IL2PD1-01/16
Record Dates: First submitted 2022-06-23; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ph I: F16IL2 + Nivolumab (Experimental): Patients will receive a fixed dose of Nivolumab and the following increasing dose levels of F16IL2: 15, 30, 50 and 70 Mio IU.
  Once the RD is established, 17 patients will receive a fixed dose of Nivolumab and F16IL2 at the RD, established during the Phase I part of the study.
  Interventions: Drug: F16IL2; Drug: Nivolumab, fixed dose

INTERVENTIONS:
Drug: F16IL2 — F16IL2 infusion will be always administered in 180 minutes i.v. on day 1, 8, 15 and 22 of each 28-days cycle.
Drug: Nivolumab, fixed dose — Patients will receive 3 mg/kg of Nivolumab as a 60 minutes i.v. infusion on day 1 and day 15 of each 28-days cycle.

SUMMARY:
Prospective, open label, non-randomized, phase I/IIb study of F16IL2 in combination with Nivolumab.

DETAILED DESCRIPTION:
The study will take place in two phases. In Phase I, the MTD and RD will be defined following a traditional 3+3 design and patients will be treated in cohorts of 3 to 6 patients with a fixed dose of Nivolumab (3 mg/kg) and escalating doses of F16IL2.

Following successful completion of the dose-finding, the study will proceed to Phase IIb and 17 patients will be treated with Nivolumab (3 mg/kg) and F16IL2 at the RD determined in Phase I.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years.
2. Subjects with histologically or cytologically-documented locally advanced NSCLC who present with stage IVA or IVB according to the 8th TNM classification. Pathological characterization must be sufficient to define patients as having either squamous or non-squamous histology.
3. Previous treatment/s for NSCLC with platinum-based 1st line therapy regimen with or without maintainance therapy and documented disease progression. First line platinum-based therapy has to consist of at least 4 cycles.
4. Patients with a known sensitizing mutation in the EGFR gene must have experienced disease progression (during or after treatment) or intolerance to treatment with afatinib, erlotinib, gefitinib, or another EGFR-TKI approved for the treatment of EGFR-mutant NSCLC. Patients with a known ALK fusion oncogene must have experienced disease progression (during or after treatment) or intolerance to treatment with crizotinib or another ALK-TKI approved for the treatment of NSCLC in patients having an ALK fusion oncogene.
5. Evaluable tumor tissue available (either FFPE tissue block or unstained tumor tissue section); fresh or archival.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
7. Patients must have at least one unidimensionally measurable lesion by computed tomography or MRIas defined by RECIST criteria 1.1.
8. Prior radiation therapy is allowed, if the irradiated area is not the only source of measurable or assessable disease and if the radiation therapy is not within 4 weeks of the administration of study treatment.
9. All acute toxic effects (excluding alopecia and fatigue) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) Grade ≤ 1.
10. All baseline laboratory requirements will be assessed and should be obtained within 21 days of treatment start. Screening laboratory values must meet the following criteria:

    * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L, platelets ≥ 100 x 109/L, haemoglobin (Hb) ≥ 9.0 g/dl.
    * Alkaline phosphatase (ALP), alanine aminotransferase (ALT) and or aspartate aminotransferase (AST) ≤ 3 x upper limit of reference range (ULN), and total bilirubin ≤ 2.0 mg/L unless liver involvement by the tumor, in which case the transaminase levels could be ≤ 5 x ULN.
    * Creatinine ≤ 1.5 ULN or creatinine clearance ≥ 30 mL/min.
11. Estimated life expectancy of at least 12 weeks.
12. Negative serum pregnancy test for females of childbearing potential*.
13. Documented negative test for HIV, HBV and HCV. For HBV serology: the determination of HBsAg, anti-HBsAg-Ab and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBsAb with no history of vaccination and/or anti-HBcAb), negative serum HBV-DNA is required. For HCV: HCV RNA or HCV antibody test. Subjects with a positive tst for HCV antibody but no detection of HCV RNA indicating no current infection are eligible.
14. Negative TB test (e.g. Mantoux or Quantiferon assay)
15. Written informed consent.

    * Subjects or legal rappresentative must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
    * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

      * Women of childbearing potential (WOCBP) must be using, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesteron-only or combined (estrogen- and progesteron-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomised partner. Pregnancy test will be repeated at the end of treatment visit.

Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilised (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion Criteria:

a. Cancer-specific exclusions

1. Any tumor therapy (chemotherapy, biologics for cancer, or an investigational therapy) within 4 weeks of the administration of study treatment.
2. Uncontrolled tumor-related pain; patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to enrollment.
3. Active symptomatic central nervous system metastases. Subjects are eligible if CNS metastases have been treated and subjects have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 4 weeks prior to the first administration of study treatment.
4. Subjects must have been either off corticosteroids, or on a stable or decreasing dose ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to enrollment.
5. Carcinomatous meningitis

   b. General Medical Exclusions
6. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study or any cancer curatively treated < 5 years prior to study entry, except cervical carcinoma in situ, non-melanoma skin cancer, superficial bladder tumors.
7. Pregnant and lactating women.
8. Uncontrolled medical condition considered as high risk for the treatment with an investigational drug (e.g. unstable diabetes mellitus, vena-cava-syndrome, uncontrolled pleural effusion, pericardial effusion).
9. Prior allogeneic bone marrow transplantation or solid organ transplant.
10. Heart failure (> Grade II, New York Heart Association Criteria - NYHA).
11. History within the last 12 months of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
12. Irreversible cardiac arrhythmias requiring permanent medication.
13. History of stroke or transient ischemic attack within the previous 12 months.
14. Severe or uncontrolled hypertension according to WHO criteria.
15. Ischemic peripheral vascular disease (Grade IIb-IV).
16. Documented history or active autoimmune disorders with the exception of:
17. skin disorders (such as vitiligo, psoriasis, or alopecia),
18. stable diabetes mellitus type 1,
19. Autoimmune thyroiditis requiring hormone replacement only.
20. Presence of primary or secondary immune deficiency.
21. Major trauma including surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
22. Known history of allergy to IL-2 or other intravenously administered human proteins/peptides/antibodies.
23. Neuropathy > Grade 2.
24. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
25. Subject unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
26. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.

    c. Exclusion criteria related to medication
27. Treatment with any investigational study drug within 4 weeks before beginning of study treatment.
28. Treatment with hematopoietic growth factors or immunomodulatory agents within 7 days of the administration of study treatment.
29. Immunosuppressive treatment within 2 weeks prior to cycle 1, day 1.
30. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to start of study drug (inhaled steroids and adrenal replacement steroid doses are permitted in absence of any active autoimmune disease)
31. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
32. Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
33. Treatment with systemic immunostimulatory agents (including but not limited to IFNs and IL-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events that are related to treatment and classified as DLTs for each administered dosage - phase I study | From Day 1 to Day 28 of treatment cycle
Objective response rate (ORR) - phase II study | At week 8
Objective response rate (ORR) - phase II study | At week 16
Objective response rate (ORR) - phase II study | At week 24

SECONDARY OUTCOMES:
Human anti-fusion protein antibodies (HAFA) levels - phase I study | 1) at day 1; 2) at day 29; 3) at day 57; 4) at day 85; 5) at day 127; 6) at day 169;
Objective response rate (ORR) - phase I study | 1) At day 52 - 56 (week 8) every 8 weeks up to 12 months; 2) At day 98 - 112 (week 16) every 8 weeks up to 12 months; 3) from week 24 every 12 weeks untils 12 months
  During treatment and after completion of administration of both Nivolumab and F16IL2 every 8 weeks up to 6 months after study initiation and then every 12 weeks until 12 months after study initiation
Progression-free survival (PFS) - phase I study | 1) At day 52 - 56 (week 8) every 8 weeks up to 12 months; 2) At day 98 - 112 (week 16) every 8 weeks up to 12 months; 3) from week 24 every 12 weeks untils 12 months
  Time from treatment start to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause
Median overall survival (mOS) - phase I study | From day 1 up to 1 year
Percentage of Participants With On-Study Adverse Events (AEs) and Serious Adverse Events (SAEs) - phase II study | From day 1 up to 1 year
Percentage of Participants With Worst On-Study Hematological and Chemistry Abnormalities - phase II study | 1) From treatment initiation to day 112 (week 16), every week; 2) At day 168 (week 24) from treatment initiation, every 12 weeks, up to 12 months
Progression-free survival (PFS) - phase II study | 1) At day 52 - 56 (week 8) every 8 weeks up to 12 months; 2) At day 98 - 112 (week 16) every 8 weeks up to 12 months; 3) from week 24 every 12 weeks untils 12 months
  Time from treatment start to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause
Median overall survival (mOS) - phase II study | From day 1 up to 1 year
Human anti-fusion protein antibodies (HAFA) levels - phase II study | 1) at day 1; 2) at day 29; 3) at day 57; 4) at day 85; 5) at day 127; 6) at day 169;

CONTACTS AND LOCATIONS:
Locations (1):
- Basel University Hospital, Basel, Switzerland